CLINICAL TRIAL: NCT06864208
Title: Piloting an Intervention to Address Weight Bias Internalization to Improve Adolescent Weight Management Outcomes
Brief Title: Addressing Weight Bias Internalization to Improve Adolescent Weight Management Outcomes: Randomized Pilot Trial
Acronym: SWIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23DK135791-02 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-02

CONDITIONS: Weight; Body Weight; Weight Bias; Weight Stigma; Physiological Stress; Biological Markers of Stress; Biological Markers of Inflammation; Eating Behaviors
Keywords: Adolescents; Teens; Weight; C-reactive protein; CRP; Interleukin-6; IL-6; Eating behaviors; Behavioral weight management; Weight bias; Weight stigma
MeSH Terms: conditions — Body Weight; Weight Prejudice; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Randomized pilot trial with active comparator
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight Bias Internalization + Behavioral Weight Management Intervention (WBI + BWM) (Experimental): WBI+BWM is a multicomponent behavioral weight loss intervention designed to address both weight bias internalization and weight status in adolescents. The first four sessions of the intervention will be focused on targeted WBI/weight stigma content, followed by 16 sessions addressing both weight stigma/WBI and evidence-based weight management strategies. Weekly meetings are scheduled for 75 minutes and are facilitated by a behavioral expert (e.g., PhD in clinical psychology). Caregivers attend 4 of the 20 weekly groups with their teens.
  Interventions: Behavioral: Behavioral Weight Management; Behavioral: Weight Bias Internalization
- Health Information Control + Behavioral Weight Management Intervention (HIC + BWM) (Active Comparator): The first four sessions (weeks 1-4) of the HIC+BWM group will focus on health promotion for adolescent health concerns other than weight management (e.g., skin cancer prevention, smoking cessation). This health information control will allow for testing of the initial 4- week WBI intervention as compared to a contact-matched control. Following the four-week health education control, the remaining 16 sessions will focus on evidence-based weight management strategies. Caregivers attend 4 of the 20 weekly groups with their teens.
  Interventions: Behavioral: Behavioral Weight Management

INTERVENTIONS:
Behavioral: Behavioral Weight Management — Prescription of diet and physical activity strategies paired with behavioral strategies for weight management
Behavioral: Weight Bias Internalization — Addressing weight stigma and improving weight-related self-perception through challenging weight-related stereotypes, practicing self-compassion, reducing self-criticism, and coping with weight stigma
  Arms: Weight Bias Internalization + Behavioral Weight Management Intervention (WBI + BWM)

SUMMARY:
Weight stigma and weight bias internalization (WBI) are common among adolescents at higher weight statuses. WBI is associated with negative physical and mental health outcomes. The current study aims to test an intervention for weight stigma and WBI combined with an evidence-based adolescent weight management program. Eligible adolescents (13-17) will be assigned by chance to one of two groups: 1) a 4-week intervention focused on weight stigma and WBI followed by a 16-week behavioral weight management program; or 2) a 4-week health information control (to include non-weight-related health promotion topics such as smoking and skin cancer prevention) followed by the same 16-week weight management program but without the WBI and weight stigma content. Study outcomes will be assessed at the 4-week and post-treatment (20 week) timepoints.

DETAILED DESCRIPTION:
The overall goal of this project is to examine the impact of intervening on weight bias internalization (WBI) in conjunction with evidence-based adolescent behavioral weight management (BWM) and to assess reduction in key mechanisms of stress resulting from weight stigma (i.e., biological markers of stress and inflammation, dysregulated eating behaviors) and subsequent impact on weight loss interference resulting from WBI.

An open trial was previously conducted to test initial acceptability and feasibility of a newly developed 20-week WBI+BWM intervention (ClinicalTrials.gov ID: NCT06389656). The intervention consisted of 4 weeks of WBI followed by a 16-week BWM intervention with integrated WBI and weight stigma content. Quantitative and qualitative feedback concerning acceptability and feasibility were solicited to refine the intervention. The current study is a randomized trial that will compare the 20-week WBI+BWM intervention developed in the open trial to a Health Information Control (HIC) + BWM condition. The HIC+BWM intervention consists of a 4-week health information control (consisting of non-weight-related health promotion topics such as smoking and skin cancer) followed by the same 16-week BMI, but without WBI and weight stigma content.

Primary and secondary outcomes will be assessed at the 4- and 20-week (post-treatment) timepoints. This study will evaluate the impact of the interventions on WBI, biological markers of stress and inflammation (cortisol, CRP, IL-6), and dysregulated eating behaviors. Changes in weight status will also be examined. Feasibility and acceptability will be measured during the pilot RCT to ensure ongoing fit of the intervention to the adolescent population. Data will provide effect size estimates of the impact on adolescent BMI for a large-scale randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Speak English;
* 13-17 years of age;
* BMI at or above >95th%ile for age and sex;
* Have at least one caregiver available to provide consent and participate in sessions;
* Agree to study participation;

Exclusion Criteria:

* Cognitive impairment or developmental delay impairing participation in a group setting;
* Current participation in a weight management program or recent weight loss of 5% of body weight or more;
* Medical condition known to impact weight or that would otherwise prevent participation;
* Current use of glucagon-like peptide-1 (GLP-1) receptor agonists;

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Total score on the Modified Weight Bias Internalization Scale (WBIS-M) | Baseline, 4-weeks post-intervention start, Post-Treatment (20 weeks)
  The validated Modified Weight Bias Internalization Scale (WBIS-M) assesses the degree to which people apply negative weight-based stereotypes to themselves and judge themselves negatively due to their weight. Total scores range from 1 to 77, with higher scores indicating a greater degree of WBI.
Total score on the Weight Self-Stigma Questionnaire (WSSQ) | Baseline, 4-weeks post-intervention start, Post-Treatment (20 weeks)
  The Weight Self-Stigma Questionnaire (WSSQ) measures weight-related self-devaluation and fear of enacted stigma. Total scores range from 12 to 60, with higher scores indicating a greater degree of internalized stigma.
Total score on the weight-related teasing sub-scale of the Perception of Teasing Scale (POTS) | Baseline, 4-weeks post-intervention start, Post-Treatment (20 weeks)
  The validated Perception of Teasing Scale (POTS) will be used to measure adolescents' experiences of weight based stigma separate from WBI. The scale has two sub-scales: a weight-related teasing sub-scale and a competency-related teasing subscale. Total scores on the weight-related teasing sub-scale range from 6-30, with higher scores indicating a higher frequency of historical weight-based teasing.
Average (AUC) for diurnal cortisol | Baseline, 4-weeks post-intervention start, Post-Treatment (20 weeks)
  Samples will be collected by teens at home over the course of 2 consecutive days following each assessment timepoint. A total of six samples will be collected with three samples each day: a sample immediately upon waking, another 30-60 minutes after waking, and a final sample at bedtime.
  Area under the curve (AUC) will be calculated for diurnal cortisol. The average AUC over the course of two days at each assessment timepoint will be used in analyses.
Concentration of c-reactive protein (CRP) | Baseline, 4-weeks post-intervention start, Post-Treatment (20 weeks)
  Circulating concentration of CRP will be determined using a high-sensitivity assay based on particle enhanced immunonephelometry.
Concentration of interleukin-6 (IL-6) | Baseline, 4-weeks post-intervention start, Post-Treatment (20 weeks)
  IL-6 concentration will be determined by specific enzyme-linked immunosorbent assay.
Dysregulated Eating Behaviors | Baseline, 4-weeks post-intervention start, Post-Treatment (20 weeks)
  Disordered eating will be measured using the 36-item Eating Disordered Examination Questionnaire.

SECONDARY OUTCOMES:
Attendance rates at intervention sessions | Post-Treatment (5 months)
  Feasibility includes the extent to which adolescents are able to utilize the intervention components offered. Attendance at group sessions will be used to measure feasibility.
Retention rate for intervention sessions | Post-Treatment (5 months)
  Feasibility includes the extent to which adolescents are able to utilize the intervention components offered. Retention, as measured by the drop-out rate for the intervention program, will be used to measure feasibility.
Total score on an adapted version of the Acceptability of Intervention Measure (AIM) | Data collected after each intervention session (20 sessions, 20 weeks)
  Intervention acceptability refers to the extent to which the WBI+BWC intervention is agreeable, palatable, or satisfactory to adolescents engaging in the treatment. We adapted the validated Acceptability of Intervention Measure (AIM) to assess adolescent acceptance related to treatment components following each intervention session. Total scores range from 10-50, with higher scores indicative of higher levels of intervention acceptability.

OTHER OUTCOMES:
Anthropometrics | Baseline, 4-weeks post-intervention start, Post-Treatment (20 weeks)
  Height will be measured in triplicate using a stationary stadiometer to the nearest 0.1 cm. Body weight will be measured in triplicate using a calibrated digital scale to the nearest 0.1 kg. The average height and weight measurements will be used to calculate body mass index (BMI) and percent of the 95th percentile of BMI for age and sex.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Darling, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes